CLINICAL TRIAL: NCT04367636
Title: The Effects of Attention Training on Emotion Regulation and Stress Related Complaints During COVID-19: Validation of a New Online Treatment
Brief Title: The Effects of Attention Training on Emotion Regulation and Stress Related Complaints During COVID-19
Acronym: OCAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to technical difficulties with the online intervention
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EC/2019/0841
Record Dates: First submitted 2020-04-20; First posted 2020-04-29 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Rumination; Anxiety; Stress; Depressive Symptoms
MeSH Terms: conditions — Rumination Syndrome; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: PSE + OCAT-sham (Active Comparator): Psycho-education video + an active placebo training, consisting of 10 sessions of ±15 minutes each (during an intervention period of two weeks), will be administered. The training task is an undirected scrambled sentences task with online contingent feedback.
  Interventions: Behavioral: Behavioral: OCAT-sham; Other: psycho-education video
- Experimental: PSE + OCAT (Experimental): Psycho-education video + an attention training, consisting of 10 sessions of ±15 minutes each (during an intervention period of two weeks), will be administered. The training task is a positively directed scrambled sentences task with online contingent feedback.
  Interventions: Behavioral: Behavioral: OCAT; Other: psycho-education video

INTERVENTIONS:
Behavioral: Behavioral: OCAT-sham — Placebo version of the online contingent attention training preceded by psycho-education movieclip.
  Arms: Active Comparator: PSE + OCAT-sham
Behavioral: Behavioral: OCAT — Online contingent attention training preceded by psycho-education movieclip.
  Arms: Experimental: PSE + OCAT
Other: psycho-education video — Both groups get to see a psycho-education video before the smartphone training starts.

SUMMARY:
Attention control for external information and cognitive control for internal information play a causal role in emotion regulation according to different theories and empirical research. Former research in the lab of the investigators has shown positive effects of an interactive attention control/interpretation training, in which participants learned to unscramble scrambled sentences ("life is my a party mess") in a positive way ("my life is a party") by getting eye-tracking feedback about attention for positive ("party") vs. negative information ("mess"). After the training, participants could better reinterpret negative photos in a positive way. Attention- and cognitive control mechanisms prior to negative stressors (proactive control) and after negative stressors (reactive control) seem to play a role in this. Moreover, research has shown that low perceived control and negative expectations about future emotion regulation skills results in lower proactive control and a higher need of reactive control. Based on this, the assumption can be made that the effects of attention control training - targeting reactive control - could benefit from adding techniques that affect proactive control (e.g. psycho-education). In the present study this is investigated by testing a new two weeks attention control training to see if this has a positive effect on stress related complaints, depressive symptoms and emotion regulation. Given that the current COVID-19 pandemic is perceived as very stressful by a lot of people, the training could help here. Participants between 18 to 65 years of age are recruited during this corona crisis. The attention control training is a new smartphone based application. Participants have to unscramble scrambled sentences into grammatically correct sentences. In the training condition, participants are asked to unscramble the scrambled sentences in a positive way. By swiping, participants can see part of the sentences. This gives the investigators an image about the processing of the sentences. This procedure allows to measure how long participants attend to positive and negative words. In the training condition participants get feedback about the duration they process positive and negative words. In the control group participants unscramble the sentences as fast as possible without feedback on emotional attention. Participants only get feedback about the speed at which sentences are unscrambled. Before and after the 10 training sessions, attention of the participants is measured to see the effects of the training. Questionnaires on depressive and anxiety complaints, emotion regulation strategies, well-being and stress are administered before and after the training. There is also a follow-up measure 2 months after the training. Both groups (training and control) watch a psycho-education video before the start of the training.

ELIGIBILITY:
Inclusion Criteria:

* Android smartphone

Exclusion Criteria:

* severe depressive complaints

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Changes in depression-, anxiety- and psychosomatic stress symptoms | pre-test (before starting the training), post-test (immediately after the training), follow-up (two months after the training)
  Measured by Mood and Anxiety Symptom Questionnaire (MASQ-30). It measures the dimensions of Clark and Watson's tripartite model, covering both shared and distinct symptoms of depression and anxiety. It has three sub-scales: Negative Affect (NA), associated with both depression and anxiety; lack of Positive Affect (PA), associated with depressive moods; and Somatic Arousal (SA), associated with anxiety. Scores are ranging from 10 to 50, with higher scores indicating more severe psychopathology.

SECONDARY OUTCOMES:
Changes in rumination. | pre-test (before starting the training), post-test (immediately after the training), follow-up (two months after the training)
  Measured by Rumination Response Scale (RRS). This 22-item questionnaire provides a total rumination score (range: 22 - 88), as well as Brooding and Reflection sub-scale scores (range: 5 - 20). Brooding is characterized by a passive style of moody pondering. Higher scores indicate a worse outcome.
Changes in cognitive emotion regulation strategies. | pre-test (before starting the training), post-test (immediately after the training), follow-up (two months after the training)
  Measured by the Cognitive Emotion Regulation Questionnaire (CERQ). Which measures different emotion regulation strategies. This questionnaire has 9 sub-scales: self-blame, other-blame, rumination, catastrophizing, putting into perspective, positive refocusing, positive reappraisal, acceptance and planning. Each sub-scale has a scoring range between 4 and 20. A higher score represents a greater frequency of engaging in that emotion regulation strategy.
Changes in emotional attention | pre-test (before starting the training), post-test (immediately after the training)
  Measured by a baseline measure in our OCAT app and measure of the end of the training period.

OTHER OUTCOMES:
How variables related to COVID-19 and the quarantine affect the life of participants | pre-test (before starting the training)
  Measured by the COVID questionnaire (designed by the researchers).
Changes in depressive complaints | pre-test (before starting the training), post-test (immediately after the training), follow-up (two months after the training)
  Measured by Center for Epidemiological Studies - Depression (CES-D), which has 20 items. A higher score represents more depressive feelings (range: 0 - 60).
Changes in symptoms of anxiety | pre-test (before starting the training), post-test (immediately after the training), follow-up (two months after the training)
  Measured by the Generalized Anxiety Disorder 7 item scale (GAD-7). Scores may vary from 0 to >15. A higher score represents more symptoms of anxiety.
Changes in well-being | pre-test (before starting the training), post-test (immediately after the training), follow-up (two months after the training)
  Measured by the Warwick-Edinburgh Mental Well-being Scales (WE-MWB). This 14-item scale indexes positive aspects of mental health. Scores may vary between 14 and 70. A higher score represents a more positive mental health.
Changes in perceived stress | pre-test (before starting the training), post-test (immediately after the training), follow-up (two months after the training)
  Measured by a Visual Analogue Stress Scale, is scored from 1 (not at all) - 10 (a lot).
Treatment Credibility and Expectancy | post-test (immediately after the training)
  Measured by the Credibility/Expectancy Questionnaire (CEQ). It measures participants' credibility and expectancy of the training. In the credibility scale the items are rated on 9- point scales ranging from 1 (Not at all logical/useful/confident) to 9 (Very logical/effective/confident). This leads to a total score on this scale between 3 and 27.
  In the expectancy scale the same 9-point scale is used and an 11-point scale (from 0% to 100%). Responses are standardized to get the total expectancy score. Higher scores represent higher credibility and expectancy.
Perceived pleasantness of the training | post-test (immediately after the training)
  A question was added to determine how pleasant the training is perceived by the participants. It is scored on a scale from 0 to 10 where 0 stands for "very unpleasant" and 10 stands for "very pleasant".

CONTACTS AND LOCATIONS:
Overall Officials: Rudi De Raedt, PhD, Principal Investigator — University Ghent; Ernst Koster, PhD, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Oost-Vlaanderen, Belgium